CLINICAL TRIAL: NCT06568406
Title: Definition of the Effect of Early Individual Physiotherapy on Evaluation of Pain, Quality of Life, Function of the Pelvic Floor Muscles, and on the Sexual Functions in Women Following an Episiotomy During a Delivery
Brief Title: Impact of Early Physiotherapy on Pain, Quality of Life, Pelvic Floor Function, and Sexual Health Post-Episiotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Ladislav Batalik, Principal Investigator, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Epi-Fyzio
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Gynecological; Surgery (Previous), Causing Obstructed Labor
Keywords: Episiotomy; physiotherapy; pelvic floor; scar; pain; dyspareunia; sexual dysfunction; quality of life
MeSH Terms: conditions — Cicatrix; Pain; Dyspareunia; Sexual Dysfunction, Physiological | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scheduled Physiotherapy (Intervention) (Experimental): The mothers in the group A will be referred to the physiotherapist's office at predetermined intervals (intervention group) compared to the current care system.
  Interventions: Procedure: Physiotherapy; Diagnostic Test: Urogynaecology
- Standard Care (Control) (Active Comparator): The mothers included in the group B will undergo standard care in the established manner at the Department of Obstetrics and Gynecology of the Faculty Hospital in Brno, which consists of routine treatment of the perineum and inspection of the perineum by a doctor that by rule occurs the 3rd day after delivery and by the end of the hospitalization
  Interventions: Diagnostic Test: Urogynaecology

INTERVENTIONS:
Procedure: Physiotherapy — Examination by a physiotherapist: the first check-up with an examination and a therapeutic intervention with the patient is performed within 24-72 hours after delivery. This is followed by two regular outpatient check-ups by a physiotherapist for the purpose of therapy and education. The second check takes place after 6-8 weeks. And the third check occurs after 10-14 weeks after childbirth. In these three checks, data collection is carried out simultaneously (in order to complete the secondary objective). The patients are examined and monitored by the same physiotherapist.
  Arms: Scheduled Physiotherapy (Intervention)
Diagnostic Test: Urogynaecology — Examination by a urogynaecologist this is carried out in the period of 14-18 weeks after childbirth in order to complete the primary objective. Data collection in order to complete the primary objective is done in the period of 14-18 weeks and 12-14 months after delivery (the online method without the need for a physical visit is preferred).

SUMMARY:
Surgical incision of the perineum and the posterior vaginal wall during a vaginal delivery (episiotomy) is among the most common surgical procedures performed in obstetrics. On the condition of having been performed correctly and in certain situations, episiotomy can be beneficial for a mother in decreasing the risk of a serious perineum injury. The benefit for a foetus can lie in acceleration of the final stage of delivery in the event of acute foetal distress. Many adverse effects are however connected to episiotomy. The morbidity connected to episiotomy can affect physical, mental, and social well-being of women during immediate as well as long-term post-partum periods. Currently, there are no universal standards that would describe and recommend physiotherapy for women following episiotomy during the first days, weeks, and months after a delivery. Care about the wound and the resulting scar after giving birth with episiotomy is an important topic because clinical experience shows that scars in the perineal area can have negative effects on the function of the pelvic floor muscles, on perineum pains, sexual health, and on mental well-being of a woman. Treatment of women with perineal wounds therefore requires a multidisciplinary approach, in which doctors, physiotherapists, and other medical professionals should be aware of the impact of a perineal scar on the quality of woman's life. Treatment or perineal scars, external genitalia, and the pelvic floor together with a targeted education of women in individual care after their scars should be part of evidence-based practice.

DETAILED DESCRIPTION:
Project Objectives Evaluate the benefits, advantages, and disadvantages of early individual physiotherapy on the selected parameters in women following a performed uncomplicated episiotomy during a vaginal delivery.

Primary objective: Specification of the differences between two groups of expectant mothers following an uncomplicated episiotomy based on the results of a survey. The comparison is carried out between a group of mothers who underwent individual postnatal physiotherapy treatment and another group of mothers that were treated in a standard way.

Secondary objective: Evaluation of the functional changes in mothers that underwent individual physiotherapeutic treatment following an uncomplicated episiotomy.

ELIGIBILITY:
Inclusion Criteria:

* female aged 18 to 40
* following an uncomplicated mediolateral episiotomy
* primipara at term with the cephalic occiput anterior position of the foetus
* signature of the informed consent and understanding of the study protocol

Exclusion Criteria:

* premature birth prior to 37+0
* other presentation than the cephalic occiput anterior position
* a performed vaginal extraction
* an associated vaginal rupture
* an injury of the anal sphincter
* paravaginal haematoma immediately after birth and before inclusion in the study
* multiple sclerosis
* serious neurological disorders
* connective tissue diseases
* chronic inflammatory bowel diseases
* congenital developmental disorders of the external genitalia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain in the perineal space | Change from baseline to 14-18 weeks and 12-14 months
  The Short-Form McGill Pain Questionnaire (SF-MPQ) is a concise tool for assessing pain, derived from the original McGill Pain Questionnaire. It consists of three components: the Pain Rating Index (PRI), which includes 15 descriptors (11 sensory and 4 affective) rated on a scale from 0 to 3; the Present Pain Intensity (PPI), where pain is rated on a 6-point scale; and, in some versions, a Visual Analog Scale (VAS), where pain intensity is marked on a 10 cm line.
Complications of healing of birth trauma | Change from baseline to 14-18 weeks and 12-14 months
  The description refers to the observation of wound complications by a physician, including the appearance of dehiscences (wound separations), secondary healing (delayed healing process), hematomas (localized collections of blood), infections in the wound, and the need for resuturing of the perineum. These complications are typically monitored post-surgery or after childbirth to ensure proper wound healing and to manage any issues that arise.
Pain in the perineum in relation to bodily and motor functions | Change from baseline to 14-18 weeks and 12-14 months
  A Visual Analog Scale (VAS) related to Activities of Daily Living (ADL) is a tool used to assess the impact of pain or other symptoms on a person's ability to perform daily tasks. The VAS typically consists of a horizontal line, usually 10 cm in length, with endpoints labeled to represent the extremes of the symptom's effect-such as "No impact on ADL" at one end and "Completely unable to perform ADL" at the other.
  Patients are asked to mark a point on the line that represents the extent to which their condition affects their daily activities. The distance from the "No impact" end to the patient's mark is measured in centimeters or millimeters, providing a quantifiable score that reflects the severity of the impact on their ability to carry out ADL. This tool is widely used in clinical settings to monitor changes over time and to evaluate the effectiveness of treatments aimed at improving functional independence.

SECONDARY OUTCOMES:
The quality of sexual functions | Change from baseline to 14-18 weeks and 12-14 months
  The Female Sexual Function Index (FSFI) is a standardized 19-item questionnaire used to assess various aspects of female sexual function, including desire, arousal, lubrication, orgasm, satisfaction, and pain. Each domain is scored separately, with higher scores indicating better sexual function, and the total score ranging from 2 to 36. The FSFI is widely used in clinical and research settings to diagnose female sexual dysfunction and monitor treatment outcomes, offering a comprehensive and validated tool for evaluating sexual health in women.
Quality of life of people with urinary incontinence | Change from baseline to 14-18 weeks and 12-14 months
  The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) is a standardized tool used to assess the severity and impact of urinary incontinence on quality of life. It consists of a few questions that evaluate the frequency, amount of leakage, and the overall impact of urinary incontinence on daily activities. Additionally, it includes a self-diagnostic item to help identify the type of incontinence. The ICIQ-UI SF is widely used in both clinical practice and research to quickly and effectively assess urinary incontinence and guide treatment decisions.
Health related quality of life | Change from baseline to 14-18 weeks and 12-14 months
  The Euro Quality of Life Five Dimensions (EQ-5D-5L) is a standardized questionnaire used to measure health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is assessed on a five-level scale, ranging from no problems to extreme problems, allowing for a detailed evaluation of a person's health status. The questionnaire also includes a Visual Analog Scale (VAS) where respondents rate their overall health on a scale from 0 to 100. The EQ-5D-5L is commonly used in clinical and research settings to assess health outcomes, inform healthcare decisions, and evaluate the effectiveness of interventions.
The functions of the pelvic floor muscles by palpation per vaginam and records them using the OXFORD SCALE | Change from baseline to 10-14 weeks
  The Oxford Scale, also known as the Medical Research Council (MRC) scale, is a tool used to assess muscle strength. It ranges from 0 to 5, with 0 indicating no muscle contraction and 5 representing normal strength with full resistance. This scale is widely used in clinical settings, particularly in neurology and rehabilitation, to evaluate and monitor muscle strength.
The functions of the pelvic floor muscles by palpation per vaginam and records them using the PERFECT SCHEME | Change from baseline to 10-14 weeks
  The PERFECT Scheme is a method for assessing pelvic floor muscle function. It stands for Power, Endurance, Repetitions, Fast contractions, Every contraction, Coordination, and Timing. This comprehensive approach is used to evaluate and treat pelvic floor disorders, such as incontinence, allowing for tailored rehabilitation and progress tracking.
The presence of possible motion synkinesis | Change from baseline to 10-14 weeks
  The physiotherapist investigates the presence of possible motion synkinesis in an attempt to activate the pelvic floor muscles - short adductors of the hips and gluteal muscles. Presence of motion synkinesis.
The condition of the wound | Change from baseline to 10-14 weeks
  The physiotherapist examines the condition of the wound and its surroundings by palpation per vaginam. They assess the presence of any swelling and haematoma of the pubic region (presence YES x NO). They assess the sensitivity (the skin sensitivity and the vaginal sensitivity: increased x decreased x no sensitivity).
The condition of the scar | Change from baseline to 10-14 weeks
  The physiotherapist checks the condition of the scar and the surrounding soft tissues of the pelvic floor by palpation per vaginam. They assess the sensitivity per vaginam using palpation (record: decreased x increased x no sensitivity), painfulness (presence YES x NO), displacement of the scar in relation to the bottom (presence YES x NO), and elastici-ty of the scars (presence YES x NO).
The presence of the abdominal separation | Change from baseline to 10-14 weeks
  The physiotherapist examines the presence of the abdominal separation (DRA). The DRA is examined using palpation. The prevalence of DRA is analyzed and recorded as YES/NO.
Hypermobility | Change from baseline to 10-14 weeks
  The physiotherapist examines hypermobility. The hypermobility is measured using the Beighton score.
  The Beighton Score is a quick assessment tool used to evaluate joint hypermobility, commonly in the context of conditions like Ehlers-Danlos Syndrome. It involves scoring five specific movements, with a total score ranging from 0 to 9. Points are awarded for hyperextension of the little fingers, thumbs, elbows, knees, and the ability to place palms flat on the floor with straight knees. A score of 4 or more suggests generalized hypermobility, while a lower score is typically considered within the normal range. This simple test helps identify individuals with hypermobility and is often part of a broader diagnostic evaluation.
Satisfaction with physiotherapy | Change from baseline to 10-14 weeks
  The physiotherapist hands the expectant woman the Likert scale to measure the satisfaction with the early physiotherapy care.
  A Likert scale is a widely used rating scale that measures attitudes, opinions, or perceptions by asking respondents to indicate their level of agreement or disagreement with a series of statements. It typically consists of 5 or 7 points, ranging from one extreme to another, such as "Strongly Disagree" to "Strongly Agree," with a neutral option in the middle (e.g., "Neither Agree nor Disagree"). The Likert scale is commonly used in surveys and questionnaires to quantify subjective data, making it easier to analyze and interpret responses in a standardized manner.

CONTACTS AND LOCATIONS:
Overall Officials: Lukáš Hruban, PhD, Principal Investigator — University Hospital Brno, Czechia
Locations (1):
- University Hospital, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No